CLINICAL TRIAL: NCT02082314
Title: Prospective Study Determining the Pain Response, Functional Interference and Quality of Life in Patients Undergoing Radiofrequency Ablation Assisted Vertebroplasty/ Cementoplasty
Acronym: RFA
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Elizabeth David, PI, Sunnybrook Health Sciences Centre
Other Study IDs: RFA
Record Dates: First submitted 2014-02-24; First posted 2014-03-10 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Neoplasms; Cementoplasty; Quality of Life
Keywords: radiofrequency ablation; bone metastases
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: RFA Vertebroplasty

SUMMARY:
Bone metastases are a cause of significant morbidity in cancer patients. In patients who die from breast, prostate, and lung cancer, autopsy studies have shown that up to 85% have evidence of bone metastases at the time of death (1). These metastases frequently give rise to complications that reduce patients' quality of life. These include: pain, fractures, and decreased mobility, ultimately reducing performance status.

Radiofrequency ablation therapy with cementoplasty/vertebroplasty for painful bone metastases has been shown to be feasible, efficacious, and safe. However, patient reported outcomes have yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven malignancy.
2. Patients aged 18 and above.
3. Advanced cancer with bone metastasis(es) to the spine and/or pelvis
4. Symptomatic with axial pain from spinal lesions and at risk for pathological fracture, or, pathological fracture without spinal cord compromise
5. Karnofsky Performance Status (KPS) greater than or equal to 40 at the time of baseline evaluation.
6. Is planned to receive RFA and/or cementoplasty with treatment to all sites being followed for study.
7. Is able to provide worst pain score at bony metastatic site(s).
8. Patient is able and willing to fill out daily diary.
9. Patients must be able to provide informed consent prior to being enrolled to the study.

Exclusion Criteria:

1. Progressive neurological compromise
2. Pathological fracture of vertebrae with significant cortical involvement or spinal canal compromise
3. Central nervous system metastases
4. Inability to record pain score, complete diary and communicate this to study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be derived from patients with advanced cancers with spinal/pelvic metastases who have been referred to interventional radiology and have consented to receiving RFA and/or cementoplasty for their disease. Such patients will be followed with a daily diary for 10 days after treatment. The Brief Pain Inventory will be used to assess pain and functional interference on these days.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain response | Baseline to 6 weeks post treatment
  To determine the complete and partial pain response rates in patients who undergo radiofrequency ablation (RFA) and/or cementoplasty/vertebroplasty for spinal/pelvic metastases.

SECONDARY OUTCOMES:
Functional Interference | Baseline - 6 weeks post treatment
  To investigate how functional interference of pain changes
Quality of Life | Baseline - 6 weeks post treatment
  To investigate quality of life changes
Side-effects | Baseline-6 weeks post treatment
  To investigate acute side effects of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth David, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No